CLINICAL TRIAL: NCT05002023
Title: PRINCE - PRenatal Identification of Childrens HEalth
Brief Title: PRINCE Study - Cohort Study of Healthy Pregnant Women Followed by the Assessment of Children´s Health and Immunity
Acronym: PRINCE
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Anke Diemert, PD Dr. med. Anke Diemert, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: PV3694
Record Dates: First submitted 2021-04-27; First posted 2021-08-12 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy; Immune System Disorder
Keywords: Pregnancy; Immune System; Birth cohort; Fetal Programming
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, white cells, cord blood, hair
Oversight: Data Monitoring Committee: Yes

SUMMARY:
In the PRINCE study we recruit healthy but also diseased pregnant women into a cohort study, followed by the assessment of children´s health and immunity at birth and during the first 10 years of life. This unique cohort allows for testing the impact of prenatal challenges on children´s health.

DETAILED DESCRIPTION:
Children´s Health is critically dependent of the prenatal well-being of the mother, and a number of observational studies have identified an impaired immunity in children upon prenatal challenges, such as stress perception, medication, nutrition or infection. However, concerted, in-depth studies assessing how such prenatal challenges may alter fetal development and subsequently children´s health in humans are largely lacking. In the present project, we address this limitation by recruiting healthy, but also diseased pregnant women into a cohort study, followed up by the assessment of children´s health and immunity at birth and during the first ten years of life.

Study participants are recruited early in the first trimester (12-15 weeks of gestation). By means of data security all participants receive a study number. Data processing into the data base (Redcap) is performed under this pseudonym.

During the first visit, the study team explains the enrollment conditions and the participants are asked to give their consent. Study visits include the documentation of clinically important conditions, sonographic examination of the fetus, assessment of mother´s height and weight as well as blood collection (21 ml) of the mother. Additionally we document any kind of medication-intake and nutrition data, and the participants are asked to fill in a psychometric questionnaire. Study visits are scheduled according to the week of gestation, i.e. around 13th, 20th (ultrasound only), 24th, 28th, 34th week. If women give birth in our clinic, we are able to collect cord blood after birth.

Blood samples are processed immediately and stored in our laboratory under Biobank-conditions.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* >18 years of age
* able to understand and sign the papers of consent
* singleton pregnancy

Exclusion Criteria: :

* <18 years of age
* unable to give consent
* multiple pregnancy
* nicotine abuse
* fetal aberration

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnancy
Study Population: The PRINCE cohort includes healthy or diseased pregnant women aged 18-45 years. Women gaining knowledge of the study from their gynecologist, in the clinic or from other participants.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-02-02 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Types of allergic diseases in childhood | 10 years follow up
  The different types of allergic diseases are assessed by a yearly questionnaire, a pediatric examination and lung function testing of the child aged 5 and 9 1/2 years, as well as analysing blood samples of the child aged 5 and 9 1/2 years. Main allergies we measure are inhalation allergens and infant food.

SECONDARY OUTCOMES:
influences during pregnancy that potentially affect children´s health | 10 years follow up
  assessed by maternal examination during pregnancy including ultrasound in every trimester
influences during pregnancy that potentially affect children´s health | 10 years follow up
  assessed by questionaire every trimester with questions about nutrition, infections, medication, stress (...)
influences during pregnancy that potentially affect children´s health | 10 years follow up
  assessed by analysing blood samples of the mother in every trimester and analysing cord blood

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Anke Diemert, MD, Principal Investigator — Department of Obstetrics and Fetal Medicine, Medical Center Hamburg-Eppendorf (UKE)
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany